CLINICAL TRIAL: NCT04498897
Title: A Randomized, Double-Blind, Placebo-Controlled Trial of Vortioxetine for Depressive Mood and Alcohol Use in Adults With Major Depressive Disorder and Alcohol Use Disorder
Brief Title: Vortioxetine for Treatment of Depressive Mood and Alcohol Use
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hanyang University Seoul Hospital (Other)
Responsible Party: Principal Investigator, Sungwon Roh, Professor, Hanyang University Seoul Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VTX-RCT
Record Dates: First submitted 2020-07-30; First posted 2020-08-05 (Actual); Last update posted 2020-08-05 (Actual); Status verified 2020-07

CONDITIONS: Depressive Disorder, Major; Alcoholism
MeSH Terms: conditions — Depressive Disorder, Major; Alcoholism | interventions — Vortioxetine; Acamprosate

STUDY DESIGN:
Intervention Model Description: A randomized, placebo-controlled study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blinded study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Test group (Active Comparator): Vortioxetine + Acamprosate
  Interventions: Drug: Vortioxetine; Drug: Acamprosate
- Placebo Group (Placebo Comparator): Placebo + Acamprosate
  Interventions: Drug: Acamprosate

INTERVENTIONS:
Drug: Vortioxetine — * Baseline: Vortioxetine 10mg (or placebo) + Acamprosate
  * First 2 weeks: Vortioxetine 5-10mg (or placebo) + Acamprosate
  * Last 6 weeks: Vortioxetine 5-20mg (or placebo) + Acamprosate
  Arms: Test group
Drug: Acamprosate — * Baseline: Vortioxetine 10mg (or placebo) + Acamprosate
  * First 2 weeks: Vortioxetine 5-10mg (or placebo) + Acamprosate
  * Last 6 weeks: Vortioxetine 5-20mg (or placebo) + Acamprosate

SUMMARY:
This is a randomized, double-blinded, placebo-controlled, multicenter study. A total of 128 subjects will be randomly assigned to a test group or placebo group in a 1:1 ratio. Subjects will receive vortioxetine (or placebo) and acamprosate for 6 weeks according to the treatment group. Four visits will be made (weeks 0, 2, 4, 8), and on visit 2-4 (weeks 2, 4, 8) compliance, depression symptoms, and alcohol craving will be assessed.

DETAILED DESCRIPTION:
Investigational product

* baseline: Vortioxetine 10mg (or placebo) qd + Acamprosate*
* First 2 weeks: Vortioxetine 5-10mg (or placebo) qd+ Acamprosate*
* Last 6 weeks: Vortioxetine 5-20mg (or placebo) qd + Acamprosate*

  * Acamprosate 666 mg bid for bodyweight < 60 kg; Acamprosate 666 mg tid for bodyweight ≥ 60 kg

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are able to understand the study and comply with all study procedures and willing to provide written informed consent prior to screening
* Male and female subjects aged 19 to 65 years old
* Diagnosed to have major depressive disorder and alcohol use disorder based on DSM(Diagnostic and Statistical Manual of Mental Disorders)-5 by two separate psychiatrists.
* MADRS(Montgomery Åsberg Depression Rating Scale) ≥ 26 at baseline

Exclusion Criteria:

* Subjects considered not safe to participate in the study (e.g. who has suicidal thoughts)
* Pregnant or breastfeeding
* Subjects with serious or unstable disease
* Clinical or laboratory signs of on-going hypothyroidism
* History of organic mental disorder, schizophrenia spectrum disorder, bipolar disorder, or substance abuse within 12 months (except for alcohol or nicotine abuse)
* Administration of antidepressant (MAOIs, SSRIs, SNRIs, TCAs) including vortioxetine and anti-craving medications (acamprosate, naltrexone) within 2 weeks from screening
* Administration of antipsychotic, anti-manic drugs, dopamine antagonists, anxiolytics (zolpidem more than 10mg, Benzodiazepine lorazepam equivalent dosage more than 2mg or used as alcohol withdrawal treatment) within 2 weeks from screening
* Administration of anti-depressant, fluoxetine, within 5 weeks from screening
* Subjects in need of an alcohol detoxification treatment
* Subjects in need of a hospitalization care

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2019-01-25 (Actual); Primary Completion 2021-04-04 (Estimated); Study Completion 2021-04-04 (Estimated)

PRIMARY OUTCOMES:
K-MADRS | From baseline for 8 weeks
  Korean-Version of the Montgomery-Asberg Depression Rating Scale

SECONDARY OUTCOMES:
OCDS-K | from baseline for 8 weeks
  Korean version of the Obsessive Compulsive Drinking Scale

CONTACTS AND LOCATIONS:
Overall Officials: Sungwon Roh, Principal Investigator — swroh@hanyang.ac.kr
Locations (1):
- Hanyang USH, Seoul, South Korea